CLINICAL TRIAL: NCT01606462
Title: Double-blind, Placebo-controlled, Randomized Study: Oxytocin and OXTR-genotypes Influence Behavioral and Neural Social Reactions
Brief Title: Oxytocin and Social Cognition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, MSc MD PhD, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OXT-071/10
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Male Volunteers
Keywords: oxytocin; social cognition; fMRI; oxytocin receptor gene
MeSH Terms: interventions — Oxytocin; lactitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): one application of 24 IU oxytocin per volunteer
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): sodium chloride solution, intranasal application, 3 puffs per nostril one application per volunteer
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — intranasal administration, 24 IU oxytocin; ; 3 puffs per nostril, each with 4 IU OXT
  Other Names: Oxytocin: Syntocinon-Spray, Novartis

SUMMARY:
The purpose of this study is to determine whether oxytocin influences memory of social stimuli and reaction to social stimuli. Furthermore the investigators explore the effect of oxytocin receptor (OXTR) polymorphism in terms of behavioral and neural responses to social stimuli.

DETAILED DESCRIPTION:
The prevailing view of OXT as a key facilitator of prosocial behaviors has been highly influenced by a plethora of studies in healthy volunteers, which demonstrated increased interpersonal trust, generosity, social learning/empathy and positively biased social stimulus processing as a result of OXT treatment. However, this interpretation is challenged by observations that OXT also promotes envy and schadenfreude (gloating), ethno-centrism (including prejudice, xenophobia, and racial bias), and defensive aggression towards outsiders.We investigate the neural correlates of emotion perception and subsequent memory effects of aversive and neutral stimuli. Tthe oxytocin effect on personal space is questioned. Additionally the effect of OXTR polymorphism regarding behavioral and neural response is explored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Current or past psychiatric disease
* Current or past physical illness
* Psychoactive medication
* Tobacco smokers
* MRI contraindication

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
neural correlates of emotion perception and subsequent memory effects of aversive and neutral stimuli | two years
  MRI data are analyzed using SPM8 (Wellcome Trust Centre for Neuroimaging, London, UK). In the first level analysis the following conditions are modeled: 'neutral: subsequently remembered', 'neutral: subsequently forgotten', 'aversive: subsequently remembered', and 'aversive: subsequently forgotten'.

SECONDARY OUTCOMES:
the effect of oxytocin receptor (OXTR) polymorphism in terms of behavioral and neural responses to social stimuli | two years
  behavioral social testing, fMRI analysis using SPM8, OXTR genotyping
The oxytocin effect on social behavior e.g. personal space is questioned | two years
  behavioral testing e.g. personal space

CONTACTS AND LOCATIONS:
Overall Officials: Rene Hurlemann, MSc MD PhD, Principal Investigator — Department of Psychiatry, University of Bonn, Germany
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

REFERENCES:
- See also: Click here for more information about the NEMO research group — http://renehurlemann.squarespace.com/welcome/